CLINICAL TRIAL: NCT02274714
Title: Dysmenorrhea in Women With Crohn's Disease and Ulcerative Colitis
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Other Study IDs: MDQ
Record Dates: First submitted 2014-10-15; First posted 2014-10-24 (Estimated); Last update posted 2017-01-23 (Estimated); Status verified 2017-01

CONDITIONS: Crohn's Disease; Ulcerative Colitis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Case (with IBD): Women aged 18-48 years with regular menstrual cycles AND with an established diagnosis of CD or UC involving the small bowel, colon or both
  Interventions: Other: Questionnaire Only
- Control (without IBD): Women aged 18-48 years with regular menstrual cycles and without a diagnosis of CD will qualify for the study
  Interventions: Other: Questionnaire Only

INTERVENTIONS:
Other: Questionnaire Only — Subjects will have an interview with a study coordinator to fill out questionnaires for the study

SUMMARY:
This case-control study will screen for dysmenorrhea and assess severity of menstrual symptoms in menstruating women with CD and UC compared with healthy age-matched controls. IBD activity will be characterized using previously validated clinical disease activity indices. General and health-related quality of life will be assessed using validated measures.

DETAILED DESCRIPTION:
Given the prior studies in IBD and corollary studies in IBS, we hypothesize that dysmenorrhea is more common in menstruating women with CD and UC than in the general population. Furthermore, we hypothesize that CD and UC activity as measured by non-invasive disease activity scores will be higher, and quality of life lower in women with both CD and UC and dysmenorrhea. As deciphering this complex relationship may avoid unnecessary testing or changes in therapy, we propose to characterize and compare the prevalence of dysmenorrhea in menstruating women with and without CD and UC. Furthermore, we will compare CD and UC activity and IBD-related quality of life in women with and without dysmenorrhea in a population of menstruating women with IBD. Lastly, we will compare general quality of life in women with and without either form of IBD and dysmenorrhea.

ELIGIBILITY:
Inclusion criteria.

* Cases: Women aged 18-48 years with regular menstrual cycles AND with an established diagnosis of CD or UC involving the small bowel, colon or both will be eligible for the study. Cases may be using oral, transdermal, or intravaginal hormonal contraception for the purpose of birth control. Regular menstrual cycles will be defined as cycles ranging from of 24 to 35 days and lasting 4 to 6 days for 3 consecutive months prior to study entry. Diagnosis of CD or UC must be made by an accredited physician on the basis of typical clinical symptoms and endoscopic, histologic, and/or radiographic findings
* Controls: Women aged 18-48 years with regular menstrual cycles and without a diagnosis of CD will qualify for the study. Controls may be using oral, transdermal or intravaginal hormonal contraception for the purpose of birth control. Regular menstrual cycles will be defined as described above. Frequency matching will be used to ensure controls are aged-matched.

Exclusion criteria include

* Inability to give written informed consent
* Pregnancy or breast feeding
* Primary or secondary amenorrhea
* Recent (within past 3 months) abdominal or gynecologic surgery
* Current or recent use (within past 3 months) of intradermal
* Injectable or intrauterine (hormonal or non-hormonal) contraception
* Less than 3 months post-partum, or post-menopausal status
* Women within 3 years of menarche will also be excluded due to the high prevalence of anovulatory cycles during this period
* Women will be excluded if they have a diagnosis of irritable bowel syndrome, or other functional bowel disorder
* Women with established endometriosis, pelvic inflammatory disease or other significant gynecologic pathology will also be excluded
* All participants with major medical issues, besides CD, as judged by the research team, will be excluded
* Major medical issues include significant disease of any organ system, such as heart failure, emphysema, or kidney failure

Ages: 18 Years to 48 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Cases: Women aged 18-48 years with regular menstrual cycles AND with an established diagnosis of CD or UC involving the small bowel, colon or both will be eligible for the study.
  Controls: Women aged 18-48 years with regular menstrual cycles and without a diagnosis of CD will qualify for the study
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2010-05; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Prevalence of Dysmenorrhea in menstruating women with and without IBD | 5 year study
  we propose to characterize and compare the prevalence of dysmenorrhea in menstruating women with and without CD and UC.

CONTACTS AND LOCATIONS:
Overall Officials: Sumona Saha, MD, MS, Principal Investigator — University of Wisconsin Hospital & Clinics
Locations (1):
- University of Wisconsin Hospital & Clinics, Madison, Wisconsin, United States